CLINICAL TRIAL: NCT02682498
Title: A Double Blind, Randomized Clinical Trial Comparing Postoperative Narcotic Usage in Patients Receiving Periarticular Liposomal Bupivicaine vs. Those Patients Receiving Standard Periarticular Joint Injections
Brief Title: Comparing Post-Op Narcotic Usage in Patients Receiving Periarticular Exparel vs. Standard Periarticular Joint Inj
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Joseph Brian Rinehart, Assistant Professor of Clinical Anesthesiology, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCIANES08
Record Dates: First submitted 2016-02-03; First posted 2016-02-15 (Estimated); Results first posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Knee Arthroplasty, Total; Liposomal Bupivicaine
MeSH Terms: interventions — Reference Standards

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EXPAREL® Bupivacaine Liposome Suspension (Active Comparator): Instead of injecting the standard joint injection for a case of total knee arthroplasty, Exparel-Liposomal Bupivicaine will be administered at the end of the surgery. A new sustained-release local anesthetic solution (Bupivacaine Liposome Injectable Suspension) will be injected into the soft tissues around the join after surgery. Exparel is a novel-composition of bupivacine in which the drug is dissolved into liposomes which release it slowly over a period of 72 hours.
  Interventions: Drug: (Bupivacaine Liposome Injectable Suspension)
- Standard periarticular joint injection (Active Comparator): A standard joint injection of 100ml (Clonidine 80 mcg, Epinephrine 0.5mg, Ketorolac 30mg, Ropivacaine 246.25mg, and Sodium Chloride 0.9% 48.45 ml) will be injected into the soft tissues around the joint after surgery.
  Interventions: Drug: Standard Preparation

INTERVENTIONS:
Drug: (Bupivacaine Liposome Injectable Suspension) — Instead of injecting the standard joint injection for a case of total knee arthroplasty, Exparel-lipsomal bupivacaine will be administered at the end of the surgery.
  Other Names: EXPAREL®
  Arms: EXPAREL® Bupivacaine Liposome Suspension
Drug: Standard Preparation — A standard joint injection of 100ml (Clonidine 80 mcg, Epinephrine 0.5mg, Ketorolac 30mg, Ropivacaine 246.25mg, and Sodium Chloride 0.9% 48.45 ml) will be injected into the soft tissues around the joint after surgery.
  Other Names: Standard Periarticular Joint Injection
  Arms: Standard periarticular joint injection

SUMMARY:
This study seeks to determine whether a new sustained-release local anesthetic solution (Exparel - Liposomal Bupivacaine) injected into the soft tissues around the joint after surgery will decrease opioid consumption and adverse events in opioid-tolerant patients presenting for total knee arthroplasty. The research hypothesis is that the Exparel (study) group will use less opioid in the first 48 hours post-operatively than the control group.

DETAILED DESCRIPTION:
Opioids have been prescribed with increasing frequency for non-acute, non-cancer pain in the last 15 years. Because of this, opioid tolerance in the general population has grown markedly, and opioid tolerant patients can be especially difficult to manage in the perioperative period. In general, they require much higher doses of opioids to obtain similar levels of pain-control compared to opioid-naïve patients and are susceptible to respiratory depression and other adverse events. This study seeks to determine whether a new sustained-release local anesthetic solution (Exparel - Liposomal Bupivacaine) injected into the soft tissues around the joint after surgery will decrease opioid consumption and adverse events in opioid-tolerant patients presenting for total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females age 18+ years old having total knee arthroplasty at UCI
* Meet at least one of the following criteria "opioid tolerant":
* Taking 50mg oral morphine equivalent or more per day
* On long-acting opioids (fentanyl pathc, oxycontin, methadone, etc.)
* Being followed by a chronic pain physician
* All subjects must be free of renal or hepatic dysfunction; defined as:
* Glomerular filtration rate >60 mL/min/1.73m^2
* AST & ALT <150, total bilirubin <1.0, INR <1.3 (if not taking anticoagulants)
* No active hepatitis, no jaundice

Control group- received standard periarticular injection Research group- receives Exparel injection

Exclusion Criteria:

* Allergy to local Anesthetic
* Pregnancy
* Nursing mothers
* Children<18 years of age
* Renal impairment (GFR<60 mL/min/1.73 m^2
* Hepatic impairment (active hepatitis, elevated AST or ALT, jaundice)
* Any history of ventricular arrhythmia or supraventricular tachycardia, or myocardial infarction within the last six months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Rinehart, M.D., Principal Investigator — University of California, Irvine
Locations (1):
- UC Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huxtable CA, Roberts LJ, Somogyi AA, MacIntyre PE. Acute pain management in opioid-tolerant patients: a growing challenge. Anaesth Intensive Care. 2011 Sep;39(5):804-23. doi: 10.1177/0310057X1103900505. PMID 21970125
- [Background] Zywiel MG, Stroh DA, Lee SY, Bonutti PM, Mont MA. Chronic opioid use prior to total knee arthroplasty. J Bone Joint Surg Am. 2011 Nov 2;93(21):1988-93. doi: 10.2106/JBJS.J.01473. PMID 22048093
- [Background] Patanwala AE, Jarzyna DL, Miller MD, Erstad BL. Comparison of opioid requirements and analgesic response in opioid-tolerant versus opioid-naive patients after total knee arthroplasty. Pharmacotherapy. 2008 Dec;28(12):1453-60. doi: 10.1592/phco.28.12.1453. PMID 19025426
- [Background] Urban MK, Ya Deau JT, Wukovits B, Lipnitsky JY. Ketamine as an adjunct to postoperative pain management in opioid tolerant patients after spinal fusions: a prospective randomized trial. HSS J. 2008 Feb;4(1):62-5. doi: 10.1007/s11420-007-9069-9. Epub 2007 Dec 19. PMID 18751864
- [Background] Cohen SM. Extended pain relief trial utilizing infiltration of Exparel((R)), a long-acting multivesicular liposome formulation of bupivacaine: a Phase IV health economic trial in adult patients undergoing open colectomy. J Pain Res. 2012;5:567-72. doi: 10.2147/JPR.S38621. Epub 2012 Nov 20. PMID 23204866
- [Background] Candiotti K. Liposomal bupivacaine: an innovative nonopioid local analgesic for the management of postsurgical pain. Pharmacotherapy. 2012 Sep;32(9 Suppl):19S-26S. doi: 10.1002/j.1875-9114.2012.01183.x. PMID 22956491
- [Background] Bergese SD, Ramamoorthy S, Patou G, Bramlett K, Gorfine SR, Candiotti KA. Efficacy profile of liposome bupivacaine, a novel formulation of bupivacaine for postsurgical analgesia. J Pain Res. 2012;5:107-16. doi: 10.2147/JPR.S30861. Epub 2012 May 1. PMID 22570563
- [Background] Chen Y, Zhang Y, Zhu YL, Fu PL. Efficacy and safety of an intra-operative intra-articular magnesium/ropivacaine injection for pain control following total knee arthroplasty. J Int Med Res. 2009 Nov-Dec;37(6):1733-41. doi: 10.1177/147323000903700609. PMID 20146871 (Retraction: PMID 23206489 J Int Med Res. 2012;40(5):2031)
- [Background] Fu P, Wu Y, Wu H, Li X, Qian Q, Zhu Y. Efficacy of intra-articular cocktail analgesic injection in total knee arthroplasty - a randomized controlled trial. Knee. 2009 Aug;16(4):280-4. doi: 10.1016/j.knee.2008.12.012. Epub 2009 Mar 18. PMID 19299145
- [Background] Richard BM, Newton P, Ott LR, Haan D, Brubaker AN, Cole PI, Ross PE, Rebelatto MC, Nelson KG. The Safety of EXPAREL (R) (Bupivacaine Liposome Injectable Suspension) Administered by Peripheral Nerve Block in Rabbits and Dogs. J Drug Deliv. 2012;2012:962101. doi: 10.1155/2012/962101. Epub 2012 Jan 17. PMID 22363842
- [Background] Richard BM, Rickert DE, Newton PE, Ott LR, Haan D, Brubaker AN, Cole PI, Ross PE, Rebelatto MC, Nelson KG. Safety Evaluation of EXPAREL (DepoFoam Bupivacaine) Administered by Repeated Subcutaneous Injection in Rabbits and Dogs: Species Comparison. J Drug Deliv. 2011;2011:467429. doi: 10.1155/2011/467429. Epub 2011 Oct 5. PMID 22013534
- [Background] Chahar P, Cummings KC 3rd. Liposomal bupivacaine: a review of a new bupivacaine formulation. J Pain Res. 2012;5:257-64. doi: 10.2147/JPR.S27894. Epub 2012 Aug 14. PMID 23049275
- [Background] Grant GJ, Barenholz Y, Bolotin EM, Bansinath M, Turndorf H, Piskoun B, Davidson EM. A novel liposomal bupivacaine formulation to produce ultralong-acting analgesia. Anesthesiology. 2004 Jul;101(1):133-7. doi: 10.1097/00000542-200407000-00021. PMID 15220782
- [Background] Grant GJ, Piskoun B, Bansinath M. Analgesic duration and kinetics of liposomal bupivacaine after subcutaneous injection in mice. Clin Exp Pharmacol Physiol. 2003 Dec;30(12):966-8. doi: 10.1111/j.1440-1681.2003.03933.x. PMID 14678238

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Periarticular Joint Injection: A standard joint injection of 100ml which contains Clonidine 80 mcg, Epinephrine 0.5mg, Ketorolac 30mg, Ropivacaine 246.25mg, and Sodium Chloride 0.9% 48.45 ml will be injected into the soft tissues around the joint after surgery.
Period: Overall Study
Arm/Group | EXPAREL® Bupivacaine Liposome Suspension | Standard Periarticular Joint Injection
Started | 18 | 20
Completed | 18 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EXPAREL® Bupivacaine Liposome Suspension | Standard Periarticular Joint Injection | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.14 (10.18) | 60 (12.83) | 60 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 11 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: 48 Hour Post-surgical Opioid Use
Description: A comparison of group means between the control group and study group with regards to 48 hour opioid use.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: morphine equivalents
Arm/Group | EXPAREL® Bupivacaine Liposome Suspension | Standard Periarticular Joint Injection
Number analyzed (Participants) | 20 | 18
morphine equivalents | 5.32 (1.72) | 5.07 (2.05)

2. Secondary Outcome: Recovery Room Opioid Use
Description: Post anesthesia care unit (recovery room) opioid use in total mg morphine IV equivalent in comparison of standard knee injection post-operatively.
Time Frame: Up to 48 hours
Population: The vast majority of the patients had been discharged by 72 hours post-op, making this outcome low-powered and not useful. Because of this we used the 48 hour pain measurement.
Measure: Median (Inter-Quartile Range); unit: Total morphine equivalents
Arm/Group | EXPAREL® Bupivacaine Liposome Suspension | Standard Periarticular Joint Injection
Number analyzed (Participants) | 20 | 18
Total morphine equivalents | 5 [0 to 10] | 5 [5 to 20]

3. Secondary Outcome: Average Daily Opioid Use During Admission
Description: Opioid use will be monitored daily from the time of admission in comparison of standard knee injection post-operatively.
Time Frame: Up to 48 hours
Population: as for outcome 2
Measure: Mean (Inter-Quartile Range); unit: Total Morphine Equivalents
Arm/Group | EXPAREL® Bupivacaine Liposome Suspension | Standard Periarticular Joint Injection
Number analyzed (Participants) | 20 | 18
Total Morphine Equivalents | 100 [0 to 150] | 103 [0 to 275]

4. Secondary Outcome: Average Daily Patient Pain Score
Description: Examining the average daily patient pain score in comparison of standard knee injection post-operatively. The measure is the Visual-Analog-Scale (VAS) for subjective pain reporting. The minimum 0 (no pain) and the maximum is 10 (worst pain imagineable). There is only one measure in the scale (i.e. there are no subscales). Lower scores on the VAS scale equate to less pain and are therefore desirable.
Time Frame: Up to 48 hours
Population: as for outcome 2
Measure: Mean (Inter-Quartile Range); unit: Visual Analog Scale Rating
Arm/Group | EXPAREL® Bupivacaine Liposome Suspension | Standard Periarticular Joint Injection
Number analyzed (Participants) | 20 | 18
Visual Analog Scale Rating | 4.75 [0 to 9.5] | 5.75 [0 to 9]

5. Secondary Outcome: Post-operative Complications
Description: Examining the post-operative complication in comparison of standard knee injection post-operatively.
Time Frame: Up to 1 month
Population: as for outcome 2
Measure: Number; unit: complications
Arm/Group | EXPAREL® Bupivacaine Liposome Suspension | Standard Periarticular Joint Injection
Number analyzed (Participants) | 18 | 20
complications | 0 | 0

ADVERSE EVENTS:
Time Frame: 10/24/13-8/18/15
Arm/Group | EXPAREL® Bupivacaine Liposome Suspension | Standard Periarticular Joint Injection
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/20
Other Adverse Events (participants affected / at risk) | 0/18 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No